CLINICAL TRIAL: NCT06603064
Title: Neuromodulation of Brain and Emotional Responses to Psychological Stress
Acronym: NUMBER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas Kraynak, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY24020114; K01MH137517 (NIH)
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Anxiety
Keywords: stress; emotion; transcranial magnetic stimulation; TMS; functional Magnetic Resonance Imaging; fMRI; neuromodulation; cardiovascular
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study will use a within-subject crossover design involving an 'active' TMS arm and a 'sham' (placebo) TMS arm. Each arm involves one visit (approx 2 hours each). Participants will complete both arms of the design.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, study staff, and the principal investigator will be blinded (masked) to participant assignment. The TMS coil to be used for this study is specifically designed to ensure participant and study staff blinding to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active then Sham (Experimental): In this arm, participants will first undergo active theta burst stimulation (cTBS) at the first visit and then undergo sham cTBS in the second visit.
  Interventions: Device: Active continuous theta burst stimulation; Device: Sham continuous theta burst stimulation
- Sham then Active (Experimental): In this arm, participants will first undergo sham theta burst stimulation (cTBS) at the first visit and then undergo active cTBS in the second visit.
  Interventions: Device: Active continuous theta burst stimulation; Device: Sham continuous theta burst stimulation

INTERVENTIONS:
Device: Active continuous theta burst stimulation — This intervention involves an active form of continuous theta burst stimulation (cTBS) that will be targeted to the dorsal anterior cingulate cortex based on neural navigation software. cTBS will be delivered in one session, lasting a few minutes, before participants complete additional testing.
Device: Sham continuous theta burst stimulation — This intervention involves an sham form of continuous theta burst stimulation (cTBS) that will be targeted to the dorsal anterior cingulate cortex based on neural navigation software. cTBS will be delivered in one session, lasting a few minutes, before participants complete additional testing.

SUMMARY:
Investigators are conducting this study to test if temporarily and non-invasively stimulating the brain will affect the emotional response to stress in healthy participants.

Participants will perform a series of tasks while completing an MRI scan. After this, participants will be randomized to undergo transcranial magnetic stimulation (TMS) at two visits, undergoing active stimulation at one visit and undergoing 'sham' stimulation at another visit. Immediately following both stimulation sessions, participants will repeat the tasks during MRI scanning.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30 to 50
2. English language proficiency (English as the primary language used in the home for the past 10 years)
3. Report that they will reside in the Pittsburgh area for at least 6 weeks, to maintain scheduling availability

Exclusion Criteria:

1. Medication Use

   1. The following medications can affect brain and cardiovascular measures being obtained in this study; thus, use of the following medications on one or more occasions in the past 14 days constitutes grounds for exclusion:

      * Antihypertensive or cardiac medications (diuretics, beta blockers, calcium channel blockers, ACE inhibitor/ARB, cardiac glycosides, central sympatholytic HTN drugs, anti-arrhythmic drugs, vasodilator drugs, other cardiac drugs)
      * Anticonvulsant medications
      * Anti-Parkinson medications
      * Protease inhibitors or other Anti-HIV medications
      * Medications for the treatment of mania, including antipsychotics
      * All other centrally active or psychotropic medications, excluding anxiolytic and antidepressant medications.
      * Insulin
      * Chemotherapy
      * Immunosuppressants and related biological agents (Imuran, methotrexate, and cyclophosphamide)
      * Prescription weight loss medications and ephedrine OTC
   2. Reported use of the following medications on a "regular" basis is grounds for exclusion. For this purpose, "regular use" is defined as reporting that the prescribed medication was taken 7 or more days in the past 14 days. Individuals who take these medications, but less frequently than 7 out of the past 14 days are not excluded:

      * Short-lasting benzodiazepines
      * Asthma oral medications
      * Asthma/allergy inhalants
      * Antidepressant medications
      * Glucocorticoids (e.g., oral prednisone, cortisol)
      * Medical marijuana
   3. The following medications can affect the CNS for 24 hours following administration; thus, reported use of the following medications within 48 hours of scanning is excluded:

      * Longer acting benzodiazepines
      * Sleep medications (e.g., trazodone)
   4. Reported use of more than 2 non-insulin medications for diabetes on a "regular" basis is grounds for exclusion. For this purpose, reported use of combination medications, involving two or more non-insulin medications for diabetes in a single pill, is counted as 2 separate medications and would be grounds for exclusion.
   5. A person who reports that he or she was once on a disallowed medication but has discontinued this medication for at least a month or longer and is otherwise eligible, is allowed to participate in the study.
2. Substance use exclusions:

   1. Anyone reporting 35 or more alcoholic drinks in the last 7 days is excluded.
   2. Anyone reporting consumption of 6 or more alcoholic drinks on 3 or more occasions in the past 7 days is excluded.
   3. Anyone reporting use of illicit drugs on 7 or more days in the past 2 weeks is excluded.
3. Medical conditions:

   1. Epilepsy or a history of seizures.
   2. Self-reported prior heart attack, stroke, bypass surgery, angioplasty, congestive heart failure, arrhythmia (cardiac rhythm problems).
   3. Severe hypertension (SBP/DBP > 160/and/or >100 mmHg)
   4. Cancer (treatment in last 12 months, allowances for non-melanoma skin cancer)
   5. Liver disease
   6. Kidney disease
   7. Type I diabetes
   8. Self-reported history of a major neurological disorder or brain injury resulting in ongoing symptoms or cognitive impairment (e.g., multiple sclerosis, cerebral palsy, major head injury)
   9. Self-reported chronic psychotic illness (schizophrenia, bipolar disorder)
   10. Lung disease requiring drug treatment (note however that asthma or allergy inhalers are not exclusionary unless they are used on a "regular basis")
4. Pregnant participants, or participants actively planning to become pregnant in the next 3 months, are excluded.
5. Those with a visual impairment that would prevent them from reading printed text or text on a computer screen, iPad, or other electronic device are excluded.
6. Those with color blindness, who may not be able to distinguish colors on some of the tasks used in this study, are excluded.
7. Those who report that they are not comfortable with undergoing MRI because of the confined space would be excluded. If individuals are interested in the study, but unsure about their comfortability with undergoing an MRI, then they would be given the option to try going into a mock MRI, which is a replica of an MRI scanner. This is meant to aid interested individuals in determining whether they are comfortable with having an MRI. If they report that they are comfortable after this experience, then they would be eligible to continue. If not, then they would be discontinued from further participation.
8. Those who use certain medical devices, implants, or other metal objects in or on the body that cannot be removed and are incompatible with use of fMRI (for example, tattooed eyeliner) are excluded. Many devices can be deemed MRI compatible with the make and model of medical device. If a participant reports a metal medical device, a letter from a medical professional with the make and model number of the device may be used to assess compatibility.
9. Those who are unable to fit into an MRI scanner (over 7ft2in tall or greater than 350lbs weight) are excluded.
10. Those who report working the night shift on a frequent basis (half or more of the hours worked in a full workday are between midnight and 8 am, and this has occurred more than 12 times during the past year) are excluded.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Dorsal anterior cingulate cortex activation to stress | 30-60 mins post-stimulation
  Blood-oxygen-level-dependent (BOLD) signal in a dorsal anterior cingulate cortex (dACC) region of interest mask extracted from the incongruent (stress) vs congruent (control) contrast.
Dorsal anterior cingulate cortex connectivity to stress | 30-60 mins post-stimulation
  Generalized psychophysiological interaction (gPPI) estimate reflecting stressor-evoked dorsal anterior cingulate cortex (dACC) functional connectivity to the anterior insula, amygdala, and periaqueductal gray.
Change in arousal during stress | 30-60 mins post-stimulation
  Rating on a modified self-assessment manikin scale (SAM) measuring subjective ratings of arousal ("To what extent do you feel calm?" 1 - very calm, 9 - very aroused) following the psychological stressor task compared to a pre-stressor baseline.
Change in valence during stress | 30-60 mins post-stimulation
  Rating on a modified self-assessment manikin scale (SAM) measuring subjective ratings of valence ("To what extent do you feel happy vs unhappy?" 1 - very unhappy, 9 - very unhappy) following the psychological stressor task compared to a pre-stressor baseline.
Change in perceived control during stress | 30-60 mins post-stimulation
  Rating on a modified self-assessment manikin scale (SAM) measuring subjective ratings of perceived control ("To what extent do you feel in control?" 1 - very little control, 9 - very much control) following the psychological stressor task compared to a pre-stressor baseline.
Systolic blood pressure response to stress | 30-60 mins post-stimulation
  The difference in systolic blood pressure (in mmHg) obtained during the psychological stress task compared to a resting pre-stressor period.
Heart rate response to stress | 30-60 mins post-stimulation
  The difference in heart rate (in beats per minute) obtained during the psychological stress task compared to a resting pre-stressor period.

SECONDARY OUTCOMES:
Dorsal anterior cingulate cortex (dACC) resting cerebral blood flow (rCBF) | 30-60 mins post-stimulation
  Cerebral blood flow (in mL/g/min) obtained at rest within a dorsal anterior cingulate cortex (dACC) region of interest.
Positive and Negative Affect Schedule - Expanded Form (PANAS-X) | 30-60 mins post-stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Kraynak, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will comply with all National Institute of Mental Health (NIMH) guidelines regarding data sharing and make use of NIMH databases.